CLINICAL TRIAL: NCT02498262
Title: Using Virtual Reality and Robotics Technologies for Vocational Evaluation, Training and Placement
Acronym: VR4VR
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of South Florida (Other)
Collaborators: Florida Department Of Education (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: Ame2_Pro00013008
Record Dates: First submitted 2015-06-25; First posted 2015-07-15 (Estimated); Last update posted 2019-07-12 (Actual); Status verified 2018-09

CONDITIONS: Autism Spectrum Disorder; Traumatic Brain Injury
Keywords: Severe Mobility and Manipulation Impairments
MeSH Terms: conditions — Autism Spectrum Disorder; Brain Injuries, Traumatic

ARMS (1):
- Virtual Reality Training System (Experimental)
  Interventions: Other: Virtual Reality System

INTERVENTIONS:
Other: Virtual Reality System — The participants will use a virtual reality system that is like a large video game and complete some job skill tasks in the virtual world video game.

SUMMARY:
Using Virtual Reality and Robotics Technologies for Vocational Evaluation, Training and Placement (VR4VR) is a project that incorporates Virtual Reality into job training to increase job opportunities for people who have physical or mental disabilities. The investigators are using Virtual Reality and robotics for job evaluation, training and placement of people with disabilities. The investigators' goal is to assess and train people in a safe, adaptable, and fun virtual environment similar to a video game.

This is an interventional study with three target populations: autism spectrum disorder, traumatic brain injury, and severe mobility and manipulation impairments. The prototype system allows for a wide range of environments with the vocational evaluator easily controlling the virtual experience, while the job seekers interact realistically.

DETAILED DESCRIPTION:
Study Procedures

If the participant takes part in this study, they will be asked to:

* Arrive at the Rehabilitation Robotics & Prosthetics Testbed (RRT) building at the times agreed to between the participant, the job coach and the key research personnel.
* Use a virtual reality system that is like a large video game with the job coach.
* Complete some skill tasks in the virtual world video game:

  * Cleaning skills such as vacuum cleaning, mopping and litter collection.
  * Loading virtual boxes into back of a virtual truck.
  * Fulfilling orders and deliveries with tangible boxes in a virtual warehouse.
  * Navigating to different checkpoints in an outdoor virtual environment.
  * Money management skills such as recognizing coin and bill amounts, counting money and giving correct amount of change to virtual customers.
  * Communicating with virtual characters.
* These tasks will take place in non-real virtual environments such as: warehouse, grocery, parking lot, and outside.
* The job coach or counselor will be with the participant just as they would in a traditional job training.
* The researchers will ask the participant questions about what they liked and disliked about the virtual reality system video game. These questions can be asked directly or via a form.
* There will be 15 minutes break times every hour and the total time will be equal to the participant's normal job coach interactions.
* The participant will be asked to participate no more than 5 hours each day, up to 15 days. Number of training days will be decided by the participant, the job coach, and the research staff.
* Data related to the time and the performance from the start to the end of each task will be recorded at the background automatically.
* Audio/visual and/or video documentation of the study may be recorded. Video and photographic recordings will be used only to aid in presenting the study for academic purposes. All information will be kept anonymous.
* Subjects' screening will be performed by the subjects' therapists beforehand, who will decide whether the subject is eligible for this study or not, based on the investigators' inclusion/exclusion requirements.
* Total Number of Participants: Up to 100 people (Up to 50 individuals with disabilities and Up to 50 healthy individuals) will take part in this study.

A $50 gift card will be given to each participant on their first training session as a thank you gift and an incentive to participate in the study.

ELIGIBILITY:
Inclusion Criteria:

The general inclusion criteria are as follows:

* Adults of 18-60 years of age
* Participants must display the capacity to understand the objectives of each of the skill tasks below, that will take place in various virtual environments.

Skill tasks:

* Cleaning skills such as vacuum cleaning, mopping and litter collection.
* Loading virtual boxes into back of a virtual truck using a haptic stick controller.
* Fulfilling orders and deliveries in a virtual warehouse with tangible boxes.
* Navigating to different checkpoints in an outdoor virtual environment.
* Money management skills such as recognizing coin and bill amounts, counting money and giving correct amount of change to virtual customers.
* Communicating with virtual characters.

Each target population will have additional inclusion criteria as follows:

Autism Inclusion Criteria:

* High, medium or low functioning with the ability to verbally communicate with the research team
* Being able to perform basic gestures such as extending arms and walking in place

Traumatic Brain Injury Inclusion Criteria:

* Participants will include individuals that have suffered a moderate to severe traumatic brain
* Participants must be deemed Rancho Los Amigos score of 7 or higher
* Being able to perform basic gestures such as extending arms and walking in place

Severe Mobility and Manipulation Impairments Inclusion Criteria:

• Persons with spinal cord injury, muscle dystrophy, multiple sclerosis or cerebral palsy

Exclusion Criteria:

The general exclusion criteria are as follows:

* Children less than 18 years of age
* Adults older than 60 years of age
* Pregnant women
* Participants unable to control a joystick
* Participants unable to verbally communicate

Each target population will have additional exclusion criteria as follows:

Autism Exclusion Criteria:

* Participants unable to control a joystick
* Participants unable to verbally communicate

Traumatic Brain Injury Exclusion Criteria:

* Participants unable to control a joystick
* Participants unable to verbally communicate

Severe Mobility and Manipulation Impairments Exclusion Criteria:

• Participants unable to control a joystick

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 100 (Estimated)
Dates: Start 2015-06 (Actual); Primary Completion 2019-12 (Estimated); Study Completion 2020-12 (Estimated)

PRIMARY OUTCOMES:
Improvement in composite score of performing the vocational tasks of shelving, cleaning, environmental awareness, loading back of a truck, money management and social skills. | Completion of the training (maximum three months)

CONTACTS AND LOCATIONS:
Overall Officials: Redwan Alqasemi, Ph.D., Study Director — University of South Florida
Locations (1):
- Rehabilitation Robotics & Prosthetics Testbed (RRT) Laboratory on the campus of the University of South Florida, Tampa, Florida, United States

REFERENCES:
- [Background] L. Bozgeyikli, E. Bozgeyikli, M. Clevenger, S. Gong, A. Raij, R. Alqasemi, S. Sundarrao, and R. Dubey, "VR4VR: Towards Vocational Rehabilitation of Individuals with Disabilities in Immersive Virtual Reality Environments," in proc. of Workshop on Virtual and Augmented Assistive Technologies (VAAT) at IEEE Virtual Reality 2014, Minneapolis, MN, April 2014.
- [Background] E. Bozgeyikli, L. Bozgeyikli, M. Clevenger, A. Raij, R. Alqasemi, S. Sundarrao, and R. Dubey, "Poster: Design and Development of a Virtual Reality System for Vocational Rehabilitation of Individuals with Disabilities," IEEE Symposium on 3D User Interfaces 2014, Minneapolis, MN, April 2014.
- [Background] L. Bozgeyikli, E. Bozgeyikli, M. Clevenger, S. Gong, A. Raij, R. Alqasemi, S. Sundarrao and R. Dubey, "Poster: A Virtual Reality System for Vocational Rehabilitation of Individuals with Disabilities," College of Engineering Research Day, Tampa, FL, November 2014.
- [Background] E. Bozgeyikli, L. Bozgeyikli, M. Clevenger, A. Raij, R. Alqasemi, and R. Dubey, "Poster: A Virtual Reality System for Vocational Rehabilitation of Individuals with Disabilities," College of Engineering Research Day, Tampa, FL, November 2013.